CLINICAL TRIAL: NCT00085683
Title: Human Herpesvirus-6 and Its Effect on the GABA/Glutamate Balance in the Cerebrospinal Fluid and in the Brain From Patients With Epilepsy
Brief Title: Herpes Virus-6 and Epilepsy
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040209; 04-N-0209
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-07

CONDITIONS: Epilepsy
Keywords: Magnetic Resonance Spectroscopy; Lumbar Puncture; Healthy Control Subjects; Mesial Temporal Sclerosis; Neuroexcitotoxicity; Seizure Disorder; Epilepsy; Healthy Volunteer; HV
MeSH Terms: conditions — Epilepsy; Hippocampal Sclerosis

SUMMARY:
This study will explore whether the human herpes virus-6 is associated with epileptic seizures. The virus may be involved in brain scarring, called mesial temporal sclerosis, which is seen in some epilepsy patients. The virus is also thought possibly to interfere with neurotransmitters - chemicals that brain cells use to communicate with each other. This study will measure levels of two of these chemicals, GABA and glutamate, which are believed to play a role in the development of seizures.

Patients with epilepsy, with or without mesial temporal sclerosis, and healthy control subjects 18 years of age and older may be eligible for this study. Control subjects may not be taking any medication on a regular basis. Epilepsy patients may take only phenytoin, carbamazepine, oxcarbazepine, lamotrigine, or levetiracetam. Candidates are screened with a physical examination and blood tests.

Participants have blood drawn and undergo magnetic resonance imaging (MRI) and lumbar puncture (spinal tap).

Blood Draw

Up to four teaspoons of blood are drawn through a needle in the arm for this study.

MRI

MRI uses a magnetic field and radio waves to produce pictures of the brain. The scanner is a metal cylinder surrounded by a strong magnetic field. During the scan, the subject lies on a bed that slides into the cylinder, wearing earplugs to muffle loud noises the machine makes when the magnetic fields are switched. The scan takes about 90 to 120 minutes, during which time the subject can communicate with the technician.

Lumbar Puncture

For this test the subject sits upright or lies on his or her side with knees curled at the chest. A local anesthetic is injected at the lower back, and a needle is inserted in the space between the bones where the cerebrospinal fluid circulates below the spinal cord. A small amount of fluid is collected through the needle. Collection of the fluid usually takes from 5 to 20 minutes.

DETAILED DESCRIPTION:
Objective: We would like to demonstrate with this study that the human herpesvirus-6 plays a role in the development of mesial temporal sclerosis (MTS) resulting in epilepsy. We would also like to examine what influence the virus has on the neurotransmitters glutamate and GABA, since we believe that an imbalance of the major excitatory and inhibitory neurotransmitters plays an important role in epilepsy.

Study population: The study population will consist of adult patients with epilepsy and MTS and adult patients with epilepsy and no MTS as confirmed on magnetic resonance (MR) imaging scan of the brain. We will compare findings in these two groups to those in healthy adult volunteers.

Design: This is a natural history study in which we will demonstrate the presence or absence of human herpesvirus-6 in the serum and cerebrospinal fluid (CSF) obtained from each of three adult study groups: patients with epilepsy and MTS, patients with epilepsy and no MTS, and normal controls. We will measure in all three groups the concentration of GABA and glutamate in CSF. In all three groups we will perform proton MR spectroscopy to non-invasively measure these metabolites in the brain.

Outcome measures: The three subject groups will be compared in terms of the presence or absence of the human herpesvirus-6 in the serum and CSF and in terms of the levels of glutamate and GABA as measured in the CSF and by magnetic resonance spectroscopy of the hippocampus and temporal lobe.

ELIGIBILITY:
Subjects of any race or ethnicity will be included in the study. Any subject who has been diagnosed with medically intractable epilepsy and is eligible for the epilepsy protocol #01-N-0139 will be evaluated for entry into this study.

INCLUSION CRITERIA:

* All patients will have a seizure disorder as documented by EEG and video-EEG. Half of the patients will have radiologically documented mesial temporal sclerosis and the other half will have a brain MRI without mesial temporal sclerosis. The patients can only be on phenytoin, carbamazepine, oxcarbazepine, lamotrigine or levetiracetam, since these anti-epileptic drugs have the least or no effect on the glutamate and GABA levels in the brain. The patients can not take any other medications.
* Healthy control subjects entering the study must be free of serious disease as determined by a standard physical and neurological examination. The control subjects can not be on any medication.
* All subjects must be able to give informed consent allowing us to use the cerebrospinal fluid and serum for research.
* All subjects will have to be able to refrain from chocolate, tea and coffee (low monoamine diet; Wood et al.1979) and alcohol during the one week before the study.
* Patients must be seizure free for 48 hours prior to the lumbar tap and the MRS.

EXCLUSION CRITERIA

Subjects will be excluded if:

* They are under the age of 18
* They are female and are pregnant
* They have a history of medical disorders which can affect the concentration of cerebral metabolites, including diabetes mellitus, renal dysfunction, hepatic dysfunction and electrolyte abnormality
* They take any medication for the normal control group
* They take any medication, with the exception of phenytoin, carbamazepine, oxcarbazepine, lamotrigine and levetiracetam for the epilepsy patients
* They have a history of psychiatric and/or mood disorders
* They have implanted devices such as pacemakers, medication pumps or defibrillators, or metal in the cranium except for the mouth, intra-cardiac lines, a history of shrapnel injury or any other condition/device that may be contraindicated or prevent the acquisition of MRI
* They have a coagulopathy that prevents them from having a lumbar puncture performed
* They have had a seizure 48 hours prior to the MRS and the lumbar tap

Subjects who cannot give informed consent allowing us to use the removed fluid for research will also be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45
Dates: Start 2004-06; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Aronica E, Yankaya B, Jansen GH, Leenstra S, van Veelen CW, Gorter JA, Troost D. Ionotropic and metabotropic glutamate receptor protein expression in glioneuronal tumours from patients with intractable epilepsy. Neuropathol Appl Neurobiol. 2001 Jun;27(3):223-37. doi: 10.1046/j.0305-1846.2001.00314.x. PMID 11489142
- [Background] Asano Y, Yoshikawa T, Kajita Y, Ogura R, Suga S, Yazaki T, Nakashima T, Yamada A, Kurata T. Fatal encephalitis/encephalopathy in primary human herpesvirus-6 infection. Arch Dis Child. 1992 Dec;67(12):1484-5. doi: 10.1136/adc.67.12.1484. PMID 1336954
- [Background] Bernasconi N, Andermann F, Arnold DL, Bernasconi A. Entorhinal cortex MRI assessment in temporal, extratemporal, and idiopathic generalized epilepsy. Epilepsia. 2003 Aug;44(8):1070-4. doi: 10.1046/j.1528-1157.2003.64802.x. PMID 12887438